CLINICAL TRIAL: NCT01630044
Title: Clinical Pilot Study to Evaluate a Non-Invasive, Neurostimulation Device for Treatment of Migraine Headache
Brief Title: Neurostimulation Device for Treatment of Migraine Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scion NeuroStim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00037089
Record Dates: First submitted 2012-06-05; First posted 2012-06-28 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Migraine Headache
Keywords: caloric vestibular stimulation
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TNM device, active treatment (Experimental): This is an active-only assessment of the experimental neuromodulation device
  Interventions: Device: TNM device

INTERVENTIONS:
Device: TNM device — Non-invasive neurostimulator, home-use treatment for up to 43 days.

SUMMARY:
This is a single-site, prospective, non-randomized and open label study to investigate the feasibility of home-use CVS for the prevention of episodic migraine headache and specifically to better understand what type of waveform to apply.

ELIGIBILITY:
Inclusion Criteria:

* A history of at least four, and not more than fourteen total monthly headache days of which between four and nine were migraine headache days. (Note: Patients were permitted continued access to migraine abortive medications and were being treated at the Duke University headache clinic.)
* A history of some responsiveness (incomplete) to at least one and a maximum of two prophylactic pharmaceutical therapies (utilized concurrently);
* The investigator must have confidence in the patient's ability to reliably complete and return the Daily Headache Diary.
* Subject must be at least 18 years of age.

Exclusion Criteria:

* Individuals who were pregnant, who had a history of cardiovascular disease, who worked night shifts or who had vestibular migraine, menstrual migraine, post-traumatic migraine, a history of unstable mood disorder or unstable anxiety, moderate or greater hearing loss or a history of traumatic brain injury.
* A history within the last six months of tobacco use, narcotic or barbiturates use or experiencing one or more analgesic rebound headaches.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of migraine headache days | Length of the study, about 71 days
  Daily Headache Diary will be used by subject. A headache day is defined as a twenty-four hour period which the subject has a headache.
Severity of each and of all headaches | Length of study, 71 days
  Daily Headache Diary will be used by subject. Subject will assign the level of pain based on an eleven-point pain measurement scale from zero (no pain) to ten (most intense pain).

SECONDARY OUTCOMES:
Total Monthly Headache Pain Score | Length of study, about 71 days
  The monthly measure would be the cumulative maximal headache pain scores for all headache days (days on which the subject's head pain level is one or higher on the pain measurement scale) during the month.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Laskowitz, MD, Principal Investigator — Duke University
Locations (1):
- Duke Medicine / Neurology, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Black RD, Rogers LL, Ade KK, Nicoletto HA, Adkins HD, Laskowitz DT. Non-Invasive Neuromodulation Using Time-Varying Caloric Vestibular Stimulation. IEEE J Transl Eng Health Med. 2016 Oct 7;4:2000310. doi: 10.1109/JTEHM.2016.2615899. eCollection 2016. PMID 27777829